CLINICAL TRIAL: NCT05408988
Title: The Relationship Between Urine Metanephrine Concentration and Myocardial and Lung Injury in Subarachnoid Haemorrhage Patients: a Prospective Observational Study
Brief Title: Neurogenic Myocardial and Lung Injury in SAH Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Other Study IDs: PCN/0022/KB/206/20
Record Dates: First submitted 2022-02-02; First posted 2022-06-07 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Injury; Lung Injury; Subarachnoid Hemorrhage
Keywords: myocardial injury; lung injury; SAH; subarachnoid haemorrhage; metanephrine; catecholamine-induced injury; Intensive Care Unit; neurocritical care
MeSH Terms: conditions — Lung Injury; Subarachnoid Hemorrhage | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with subarachnoid haemorrhage: Patients aged 18 or older hospitalized in the Intensive Care Unit with Subarachnoid Haemorrhage.
  Interventions: Diagnostic Test: hs-TnT (high-sensitive cardiac troponin T) plasma concentration; Diagnostic Test: CK-MB (creatine kinase myocardial band) plasma concentration; Diagnostic Test: CPK (creatine phosphokinase) plasma concentration; Diagnostic Test: NT-proBNP (N-terminal prohormone of brain natriuretic peptide) plasma concentration; Diagnostic Test: Metanephrine concentration in urine

INTERVENTIONS:
Diagnostic Test: hs-TnT (high-sensitive cardiac troponin T) plasma concentration — hs-TnT plasma concentration measured once every 12 hours
Diagnostic Test: CK-MB (creatine kinase myocardial band) plasma concentration — CK-MB plasma concentration measured every 12 hours
Diagnostic Test: CPK (creatine phosphokinase) plasma concentration — CPK plasma concentration measured every 12 hours
Diagnostic Test: NT-proBNP (N-terminal prohormone of brain natriuretic peptide) plasma concentration — NT-proBNP plasma concentration measured every 12 hours
Diagnostic Test: Metanephrine concentration in urine — Metanephrine concentration measured in 12-hour urine collection using spectrophotometry.

SUMMARY:
Up to this day, little is known whether the extent of brain damage in patients with SAH correlates with the degree neurogenic myocardial injury and neurogenic lung injury.

This is a prospective observational study designed to asses relationship between catecholamine surge and development of myocardial and lung injury in subarachnoid haemorrhage patients.

DETAILED DESCRIPTION:
Multiple forms of brain damage, primarily, subarachnoid haemorrhage (SAH) are frequently accompanied by neurogenic myocardial injury with changes in the electrocardiogram, accompanied by the release of markers of myocardial injury. This form of cardiac dysfunction is thought to be mediated by cellular toxicity associated with catecholamine release. Central nervous system damage in the course of intracranial haemorrhage may, in a similar pathogenic pathway, lead to neurogenic lung injury. Up to this day, little is known whether the extent of brain damage in patients with SAH correlates with the degree of neurogenic myocardial injury. Moreover, it remains unknown what is the full clinical picture and duration of this type of myocardial injury and how often it co-occurs with neurogenic lung injury. Such analysis is a fundamental and most important step in optimising the treatment of these patients.

Methods: In this prospective observational study the authors aim to recruit 30 patients with subarachnoid haemorrhage, requiring hospitalization in the Intensive Care Unit. The patients will be monitored for elevation in cardiac damage markers (hs-TnT, CPK, CK-MB, NT-proBNP) and worsening of respiratory conditions, defined by need for more invasive ventilation parameters, and subsequent changes in arterial blood gas. The above mentioned parameters will be assessed every 12 hours. Additionally, the patients will be screened for an elevation in catecholamine metabolite (metanephrine) concentration in 12-hour urine collection.

Hypothesis to be tested: Myocardial and lung injury in SAH patients is timely-associated with an increase in metanephrine concentration in urine.

ELIGIBILITY:
Inclusion Criteria:

* patients with subarachnoid haemorrhage (both aneurysmal and non-aneurysmal) with acute consciousness disturbances (Glasgow Coma Scale < 8 pts) requiring intubation and mechanical ventilation, hospitalized in the ICU for over 24 hours

Exclusion Criteria:

* severe prior pulmonary diseases
* severe prior cardiac diseases
* death in the first 72 hours of ICU stay
* need for any extracorporeal life-saving techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subarachnoid haemorrhage admitted to the Intensive Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-22 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital death (number of patients) | 7 days
  Death of the patient during the first 7 days of hospitalization.
Number of Patients with elevation in hs-TnT levels | 7 days
  hs-TnT treated as myocardial injury biomarker
Number of Patients with elevation in NT-proBNP levels | 7 days
  NT-proBNP treated as myocardial injury biomarker
Number of Patients with elevation in creatine kinase levels | 7 days
  Creatine kinase treated as myocardial injury biomarker
Number of Patients with elevation in creatine kinase MB levels | 7 days
  Creatine kinase MB treated as myocardial injury biomarker
Number of Patients with a decrease in Horowitz index | 7 days
  The decrease in Horowitz index treated as a sign of need for more invasive ventilation parameters with subsequent blood gas changes
Number of Patients with need of increased FiO2 | 7 days
  Need of increased FiO2 treated as a sign of need for more invasive ventilation parameters with subsequent blood gas changes
Number of Patients with need of increased PEEP values | 7 days
  Need of increased PEEP values treated as a sign of need for more invasive ventilation parameters with subsequent blood gas changes
Number of Patients with need for the use of neuro-muscular blocking agents | 7 days
  Need for the use of neuro-muscular blocking agents treated as a sign of need for more invasive ventilation parameters with subsequent blood gas changes

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Krzych, PhD, Study Chair — University Clinical Center prof. K. Gibiński of the Medical University of Silesia in Katowice
Locations (1):
- University Clinical Center prof. K. Gibiński of the Medical University of Silesia in Katowice, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osgood ML. Aneurysmal Subarachnoid Hemorrhage: Review of the Pathophysiology and Management Strategies. Curr Neurol Neurosci Rep. 2021 Jul 26;21(9):50. doi: 10.1007/s11910-021-01136-9. PMID 34308493
- [Background] Hofman M, Hajder N, Duda I, Krzych LJ. A Questionnaire Survey of Management of Patients with Aneurysmal Subarachnoid Haemorrhage in Poland. Int J Environ Res Public Health. 2020 Jun 11;17(11):4161. doi: 10.3390/ijerph17114161. PMID 32545225
- [Background] Wybraniec MT, Mizia-Stec K, Krzych L. Neurocardiogenic injury in subarachnoid hemorrhage: A wide spectrum of catecholamin-mediated brain-heart interactions. Cardiol J. 2014;21(3):220-8. doi: 10.5603/CJ.a2014.0019. Epub 2014 Feb 14. PMID 24526502
- [Background] Wybraniec M, Mizia-Stec K, Krzych L. Stress cardiomyopathy: yet another type of neurocardiogenic injury: 'stress cardiomyopathy'. Cardiovasc Pathol. 2014 May-Jun;23(3):113-20. doi: 10.1016/j.carpath.2013.12.003. Epub 2013 Dec 27. PMID 24462197
- [Background] Veeravagu A, Chen YR, Ludwig C, Rincon F, Maltenfort M, Jallo J, Choudhri O, Steinberg GK, Ratliff JK. Acute lung injury in patients with subarachnoid hemorrhage: a nationwide inpatient sample study. World Neurosurg. 2014 Jul-Aug;82(1-2):e235-41. doi: 10.1016/j.wneu.2014.02.030. Epub 2014 Feb 20. PMID 24560705
- [Background] Mazeraud A, Robba C, Rebora P, Iaquaniello C, Vargiolu A, Rass V, Bogossian EG, Helbok R, Taccone FS, Citerio G. Acute Distress Respiratory Syndrome After Subarachnoid Hemorrhage: Incidence and Impact on the Outcome in a Large Multicenter, Retrospective Cohort. Neurocrit Care. 2021 Jun;34(3):1000-1008. doi: 10.1007/s12028-020-01115-x. Epub 2020 Oct 20. PMID 33083966
- [Background] Anetsberger A, Jungwirth B, Blobner M, Ringel F, Bernlochner I, Heim M, Bogdanski R, Wostrack M, Schneider G, Meyer B, Graessner M, Baumgart L, Gempt J. Association of Troponin T levels and functional outcome 3 months after subarachnoid hemorrhage. Sci Rep. 2021 Aug 9;11(1):16154. doi: 10.1038/s41598-021-95717-w. PMID 34373566